CLINICAL TRIAL: NCT00958074
Title: A Phase II Prospective Non-Randomized Clinical Trial of Dose-Adjusted Schedule of Vorinostat in Patients With Primary Cutaneous T-Cell Lymphoma Who Did Not Receive Prior Systemic Therapy or Have Been Treated With Single Agent Targretin
Brief Title: Vorinostat in Patients With Primary Cutaneous T-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrei Shustov, Principal Investigator, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6914; NCI-2009-01231 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-08-10; First posted 2009-08-13 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Cutaneous T-cell Lymphoma Stage I; Cutaneous T-cell Lymphoma Stage II; Cutaneous T-cell Lymphoma Stage III; Cutaneous T-cell Lymphoma Stage IV
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Vorinostat; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort I (>=65 years old) (Experimental): 200 mg vorinostat PO QD on days 1-28. Treatment repeats every 28 days for 6 courses. Dose escalation by 100mg per day increments to maximum dose of 500mg per day in the absence of dose limiting toxicity.
  Interventions: Drug: vorinostat; Other: flow cytometry; Other: laboratory biomarker analysis
- Cohort II (<65 years old) (Experimental): 400 mg vorinostat PO QD on days 1-28. Treatment repeats every 28 days for 6 courses. Dose escalation by 100mg per day increments to maximum dose of 500mg per day in the absence of dose limiting toxicity.
  Interventions: Drug: vorinostat; Other: flow cytometry; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: flow cytometry — correlative study
Other: laboratory biomarker analysis — correlative study

SUMMARY:
This phase II trial studies the side effects and how well vorinostat works in treating patients with primary cutaneous T-cell lymphoma. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate to treatment with dose-adjusted Vorinostat schedule in subjects with cutaneous T-cell lymphoma (CTCL) who did not receive prior systematic therapy or have been treated with single agent targretin (bexarotene).

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of dose-adjusted Vorinostat schedule when administered to patients with primary cutaneous T-cell lymphoma who did not receive prior systematic therapy or have been treated with single agent targretin.

II. To determine the time to objective response in subjects with CTCL treated with dose-adjusted schedule of Vorinostat as primary therapy.

III To determine the duration of objective response in subjects with CTCL.

IV. To determine the time to loss of objective response.

V. To determine the objective response rate of extracutaneous manifestations of CTCL (lymph node enlargement, Sezary cells in peripheral blood).

VI. To compare the efficacy, toxicity and tolerability of dose-adjusted schedule to currently recommended flat dose of Vorinostat in subjects with CTCL.

OUTLINE: Patients are assigned to 1 of 2 treatment arms according to age (< 65 vs >= 65 years old).

COHORT I (>= 65 years old): Patients receive 200 mg vorinostat orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

COHORT II (< 65 years old): Patients receive 400 mg vorinostat PO QD on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females
* Histologically confirmed diagnosis of CTCL, including mycosis fungoides and/or Sezary syndrome
* Documentation of diagnosis by histologic examination should be available
* Subjects with CTCL stages IB, IIA, IIB, III, or IVA who have not received any prior systemic therapies
* Anticipated life expectancy greater than 6 months
* Performance status 0, 1, or 2 by Eastern Cooperative Oncology Group (ECOG) criteria
* Written informed consent to participate in the study
* Absolute neutrophil count (ANC) >= 1,000/mcL
* Platelets >= 75,000/mcL
* Hemoglobin >= 9 g/dL
* Prothrombin time or international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) =< 1.2 times the ULN unless the patient is receiving therapeutic anticoagulation
* Serum creatinine =< 1.5 X ULN OR calculated creatinine clearance >= 60 mL/min for patients with creatinine levels > 1.5 X institutional ULN; creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 2 X ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic aminotransaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic aminotransaminase [SGPT]) =< 3.0 X ULN
* Alkaline Phosphatase (liver fraction) =< 3.0 X ULN

Exclusion Criteria:

* Proven or suspected extracutaneous visceral CTCL involvement (M1) (CTCL stage IVB)
* Presence of lymphadenopathy is permitted
* ECOG performance status > 2
* Concomitant use of any anti-cancer therapy or immune modifier
* Concomitant use of any investigational agent or device
* Concomitant therapy with any other anti-CTCL therapy, or radiation therapy (topical corticosteroids or low dose oral corticosteroids [=< 10 mg/day prednisone or equivalent] will not be excluded, but if used, the dose and schedule must be stable during the two weeks immediately prior to study entry)
* Use of any previous systemic therapy (except single agent targretin), total skin electron beam (TSEB) therapy or extracorporeal photopheresis
* Evidence of clinically significant (uncontrolled) hypo- or hyperthyroidism
* Poorly controlled diabetes mellitus as evidenced by hemoglobin (Hgb)A1c > 6.5 mg/dl
* Recent (in the past 6 months) medically significant cardiac event (i.e. myocardial infarction, cardiac surgery)
* Presence of congestive heart failure (New York Heart Association [NYHA] class IV) or angina (NYHA class IV) or presence of a medically significant arrhythmia
* Congenital long QT syndrome
* Corrected QT interval > 480 msec on screening electrocardiogram (ECG)
* Presence of uncontrolled hypertension manifested by systolic blood pressure >= 180 mmHg and/or diastolic blood pressure >= 100 mmHg
* Documented current active infection with human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, and/or cytomegalovirus (CMV)
* Presence of uncontrolled bacterial or viral infection (subject may be receiving chronic antimicrobial therapy)
* History of culture-documented bacteremia in the previous 2 weeks
* Concurrent therapy with any histone deacetylase (HDAC)-like compound; patients treated with valproic acid for epilepsy may enroll after a 30 day washout period
* Recent change (in the past 2 weeks) in the doses or regimens of medication used for any chronic non-oncologic conditions for reasons of worsening of chronic illness (change in doses of chronic medications associated with improvement in a chronic illness are not exclusion criteria)
* Presence of any acute or chronic non-oncologic disease which, in the opinion of the investigator, is medically uncontrolled
* History of a prior malignancy with the exception of cervical intraepithelial neoplasia; non-melanoma skin cancer; adequately treated localized prostate carcinoma with prostate specific antigen (PSA) < 1.0; or who has undergone potentially curative therapy with no evidence of that disease for five years, and/or who is deemed at low risk for recurrence (< 30% probability) by his/her treating physician
* Patient with a "currently active" second malignancy, other than nonmelanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled
* Any significant medical or psychiatric condition that, in the opinion of the investigator, might prevent the subject from complying with all required study procedures
* Women of childbearing potential must have a pregnancy test within 28 days prior to registration, and must use an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 3 months after the study
* Females of childbearing potential and sexually active males, if indicated, must be willing and able to use two methods of contraception that are adequate to prevent or minimize risk of pregnancy for the duration of the study; one of which must be a barrier method
* Patient has symptomatic ascites or pleural effusion (a patient who is clinically stable following treatment for these conditions is eligible)
* Patient has had allogeneic transplant
* Patient has a history of a gastrointestinal surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Shustov, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Started | 4 | 7
Completed | 4 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old) | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 7 | 7
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Defined as either no evidence of clinical disease or marked improvement (>= 50%) decrease in the modified Severity-Weighted Assessment Tool (mSWAT) skin assessment score compared to baseline.
Time Frame: After at least 14 days. With Confirmation after additional 28 days.
Population: In cohort 1, only 3 of the 4 subjects consented were used for analysis. 1 patient in this cohort only completed 3 days of treatment before removing themselves from treatment and withdrawing consent. This patient was deemed inevaluable, as the timeframe for initial evaluation is 14 days.
Measure: Number; unit: percentage of total
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Number analyzed (Participants) | 3 | 7
percentage of total | 0 | 57

2. Secondary Outcome: Objective Response Rate of Extracutaneous Manifestations of CTCL (Lymph Node Enlargement, Sezary Cells in Peripheral Blood);
Description: Assessed by changes in the sum of the products in the greatest diameters of enlarged lymph nodes by serial computed tomography (CT) or positron emission tomography (PET)/CT scans.
Time Frame: Up to 30 days post-treatment
Population: 7 subjects with nodal disease (2 subjects >=65 and 5 subjects <= 65: 1 not evaluable)
Measure: Number; unit: participants
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Number analyzed (Participants) | 2 | 4
participants
  Overall Response | 0 | 0
  Stable Disease | 2 | 3
  Progressive Disease | 0 | 1

3. Secondary Outcome: Occurrences of Dose Adjustment as Measured by Safety/Toxicity
Description: Toxicities will be graded in severity according to the guidelines outlined in the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0.
Time Frame: Up to 30 days post-treatment
Population: 4 subjects >= 65, 7 subjects <= 65 who received at least one dose of drug.
Measure: Number; unit: Occurrences
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Number analyzed (Participants) | 4 | 7
Occurrences
  Dose delay | 1 | 2
  Dose reduction | 1 | 1
  Treatment discontinuation | 1 | 0

4. Secondary Outcome: Number of Participants With Overall Response as Measured by Sezary Cell Count
Description: Overall response defined by a clinically significant decrease in Sezary cell count (>50% decrease from baseline).
Time Frame: Baseline to 30 days post-treatment
Measure: Number; unit: participants
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Number analyzed (Participants) | 2 | 4
participants
  Overall response | 2 | 1
  Stable disease | 0 | 3

5. Secondary Outcome: Changes in the Physicians Serial Assessment of Erythroderma Score
Time Frame: Baseline to 30 days post-treatment
Population: 2 subjects >= 65, 3 subjects <= 65 with baseline erythroderma score.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Number analyzed (Participants) | 2 | 3
Participants
  No change | 2 | 0
  Reduction | 0 | 3
  Resolution | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of signing consent until 30 days after the last dose of study drug treatment administered or until any treatment related AE or laboratory abnormality resolved or stabilized.
Arm/Group | Cohort I (>=65 Years Old) | Cohort II (<65 Years Old)
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/7
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (>=65 Years Old) (N=4) | Cohort II (<65 Years Old) (N=7)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (>=65 Years Old) (N=4) | Cohort II (<65 Years Old) (N=7)
ABRASION (General disorders) | 1 (1) | 0 (0)
ANOREXIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
CHEST PAIN (Cardiac disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 6 (6)
DIZZINESS (General disorders) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ECCHYMOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ELEVATED CREATININE (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
ELEVATED GLUCOSE (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
FALL (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 2 (2) | 5 (5)
FOOT PAIN (FOOT TENDERNESS) (General disorders) | 1 (1) | 1 (1)
HAIR LOSS (ALOPECIA) (General disorders) | 0 (0) | 2 (2)
HEADACHE (General disorders) | 0 (0) | 1 (1)
HEARING LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARTBURN (Gastrointestinal disorders) | 0 (0) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTENSION (Cardiac disorders) | 0 (0) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
INSOMNIA (General disorders) | 0 (0) | 1 (1)
ITCHING/ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LOWER EXTREMITY EDEMA (Cardiac disorders) | 1 (1) | 1 (1)
MUSCOLOSKELETAL PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OCULAR INFECTION (Eye disorders) | 0 (0) | 1 (1)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2)
SCALP PAIN (General disorders) | 1 (1) | 0 (0)
SKIN CRACKING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN SHEDDING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN THICKENING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TASTE CHANGE (Dysgeusia) (Gastrointestinal disorders) | 1 (1) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
TREMORS (General disorders) | 0 (0) | 1 (1)
ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
WEIGHT LOSS (ANOREXIA) (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less